CLINICAL TRIAL: NCT05588050
Title: Validity and Reliability of Two Methods for Assessing Knee Joint Position Sense in Patients With Patellofemoral Pain Syndrome
Brief Title: Validity and Reliability of Two Methods for Assessing Knee Joint Position Sense
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, nada magdy saad el deen, assistant lecturer, Cairo University
Other Study IDs: P.T.REC/012/003957
Record Dates: First submitted 2022-10-13; First posted 2022-10-20 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral pain syndrme
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: smart phone application and AutoCAD software — to assess the validity and reliability of smart phone application and AutoCAD software in assessing knee joint position sense in patients with patellofemoral pain syndrome

SUMMARY:
The participants will be prepared for image-capture data collection by putting four squared markers, each 4 cm in diameter, will be attached to their leg at three locations while the subject in this position: (1) proximal to a quarter of the distance along a line joining the greater trochanter to the lateral knee joint line, (2) over the neck of the fibula, (3) over the proximal part of the lateral malleolus. A fourth marker will be attached over the iliotibial tract adjacent to the superior border of the patella when the subject in a sitting position.

Each participant will seat on the end of an orthopedic assessment plinth and blindfolded .

Each subject will be asked to extend his/her leg and make two angles arbitrarily from the resting position (90º) to the full extension. Photos will be taken, while they keep their leg at each position for five seconds.The bubble inclinometer will be attached to the patient leg at the resting position 90 º knee flexion.

The tested leg will be passively moved by the researcher through 20° to 60° of knee extension from a starting knee angle of 90° to a target angle which will be measured by the bubble inclinometer , the participant then actively held the leg in this position for 5 second.

A photograph of the leg in the target position will be taken using the camera which will be positioned 185 cm from the subject and 65 cm from the ground The leg will then be passively returned to the starting angle, and the participant will be instructed to actively move that leg to the target angle and hold it in this position another photograph will be taken, and the participant will be instructed to move the leg back to the starting position , the process will be repeated 3 times for each target angle with rest time 5 seconds between shots.

After completing the procedure for all subjects, the test and replicated angles will be measured using the AutoCAD software and determine the center of the markers.

Also , same angles will be measured via clinometer smart phone application in those patients to assess its validityand reliability where the participant will hold the leg for five seconds for each angle where this process will be reapeated for three times for each angle.

DETAILED DESCRIPTION:
The participants will be prepared for image-capture data collection by putting four squared markers, each 4 cm in diameter, will be attached to their leg at three locations while the subject in this position: (1) proximal to a quarter of the distance along a line joining the greater trochanter to the lateral knee joint line, (2) over the neck of the fibula, (3) over the proximal part of the lateral malleolus. A fourth marker will be attached over the iliotibial tract adjacent to the superior border of the patella when the subject in a sitting position.

Each participant will seat on the end of an orthopedic assessment plinth and blindfolded .

Each subject will be asked to extend his/her leg and make two angles arbitrarily from the resting position (90º) to the full extension. Photos will be taken, while they keep their leg at each position for five seconds.The bubble inclinometer will be attached to the patient leg at the resting position 90 º knee flexion.

The tested leg will be passively moved by the researcher through 20° to 60° of knee extension from a starting knee angle of 90° to a target angle which will be measured by the bubble inclinometer , the participant then actively held the leg in this position for 5 second.

A photograph of the leg in the target position will be taken using the camera which will be positioned 185 cm from the subject and 65 cm from the ground The leg will then be passively returned to the starting angle, and the participant will be instructed to actively move that leg to the target angle and hold it in this position another photograph will be taken, and the participant will be instructed to move the leg back to the starting position , the process will be repeated 3 times for each target angle with rest time 5 seconds between shots.

After completing the procedure for all subjects, the test and replicated angles will be measured using the AutoCAD software and determine the center of the markers.

Also , same angles will be measured via clinometer smart phone application in those patients to assess its validityand reliability where the participant will hold the leg for five seconds for each angle where this process will be reapeated for three times for each angle.

ELIGIBILITY:
Inclusion Criteria:

* 1) Anterior or retropatellar knee pain from at least 2 of the following Activities : (1) prolonged sitting; (2) stair climbing; (3) squatting; (4) running; (5) kneeling; and (6) hopping/jumping.

  2) Insidious onset of symptoms unrelated to a traumatic incident.

  3) Age of the subject 18-35 years to limit the possibility that PFPS over age 35 may have been complicated by arthritic changes, and also the subjects should have closed epiphyseal growth plates.

  4) Patient with chronic PFPS (pain > 3 months)

Exclusion Criteria:

1. Meniscal or other intraarticular pathologic conditions; cruciate or collateral ligament involvement.
2. A history of traumatic patellar subluxation or dislocation.
3. Previous surgery in the knee, ankle and hip joints.
4. Knee, ankle and hip joints osteoarthritis.
5. athletes aren't included .

   -

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: 1. Anterior or retropatellar knee pain from at least 2 of the following Activities : (1) prolonged sitting; (2) stair climbing; (3) squatting; (4) running; (5) kneeling; and (6) hopping/jumping.
  2. Insidious onset of symptoms unrelated to a traumatic incident.
  3. Age of the subject 18-35 years to limit the possibility that PFPS over age 35 may have been complicated by arthritic changes, and also the subjects should have closed epiphyseal growth plates.
  4. Patient with chronic PFPS (pain > 3 months
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
joint position sense in patients with patellofemoral pain syndrome | 2 years
  joint position sense assessment in patients with patellofemoral pain syndrome

CONTACTS AND LOCATIONS:
Overall Officials: mohamed A abdelfatah, Phd, Study Director — lecturer of orthopedic at faculty of physical therapy - cairo university
Locations (1):
- faculty of physical therapy- Cairo university, Cairo, Egypt

REFERENCES:
- [Result] Coelho VK, Gomes BSQ, Lopes TJA, Correa LA, Telles GF, Nogueira LAC. Knee proprioceptive function and physical performance of patients with patellofemoral pain: A matched case-control study. Knee. 2021 Dec;33:49-57. doi: 10.1016/j.knee.2021.08.031. Epub 2021 Sep 17. PMID 34543992